CLINICAL TRIAL: NCT03480919
Title: Shen Men Acupuncture for Anxiety Preceding Lumbar Epidural Injections in Acupuncture-naive Patients: a Randomized Controlled Trial
Brief Title: Acupuncture for Pre-Procedure Anxiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited resources
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-1525
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Results first posted 2019-10-01 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Injections, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Shen Men acupuncture (Experimental): Single acupuncture needles will be placed bilaterally onto the patient's Shen Men acupuncture point in the ear for a duration of 20 minutes.
  Interventions: Device: Shen Men acupuncture; Procedure: Epidural injection
- Sham acupuncture (Sham Comparator): Single acupuncture needles will be placed bilaterally onto a sham location in the ear for a duration of 20 minutes.
  Interventions: Procedure: Epidural injection
- Simulated acupuncture (Placebo Comparator): Acupuncture will be simulated with a paper clip.
  Interventions: Procedure: Epidural injection

INTERVENTIONS:
Device: Shen Men acupuncture — 20-minute acupuncture session
  Arms: Shen Men acupuncture
Procedure: Epidural injection — Epidural injection for the relief of back pain

SUMMARY:
It is common for patients undergoing spinal injections to report anxiety prior to the injection. Although sedation, general anesthesia, and medications can be used to reduce anxiety, the use of sedative agents during the procedure can increase the risk of spinal cord injury. The purpose of this study is to see if receiving acupuncture before a spinal injection can effectively reduce patients' anxiety. Only patients who are scheduled to receive a spinal injection at this institution will be eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Spine pathology that meets criteria for lumbar epidural injection

Exclusion Criteria:

* Unable to provide consent
* Contraindications to acupuncture (e.g., rash, skin infection, sensory loss in ear)
* Previous experience of acupuncture
* Age <18
* Pregnant women
* Non-English or Non-Spanish speaking

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shen Men Acupuncture | Sham Acupuncture | Simulated Acupuncture
Started | 1 | 2 | 1
Completed | 1 | 2 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shen Men Acupuncture | Sham Acupuncture | Simulated Acupuncture | Total
Number analyzed (Participants) | 1 | 2 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 1
  >=65 years | 0 | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (0) | 65 (0) | 87 (0) | 63 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Anxiety
Description: Change in anxiety from baseline (pre-acupuncture intervention) will be measured using the State subscale of the State Trait Anxiety Inventory (STAI). The STAI is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI is one of the first tests to assess both state and trait anxiety separately. Each type of anxiety has its own scale of 20 different questions that are scored. Scores range from 20 to 80, with higher scores correlating with greater anxiety. Low scores indicate a mild form of anxiety whereas median scores indicate a moderate form of anxiety and high scores indicate a severe form of anxiety. The 4-point scale for S-anxiety is as follows: 1.) not at all, 2.) somewhat, 3.) moderately so, 4.) very much so. The 4-point scale for T-anxiety is as follows: 1.) almost never, 2.) sometimes, 3.) often, 4.) almost always.
Time Frame: Up to 30 min post-acupuncture intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Shen Men Acupuncture | Sham Acupuncture | Simulated Acupuncture
Number analyzed (Participants) | 1 | 2 | 1
score on a scale | 0 (0) | 0.2 (4.5) | -6 (0)

2. Secondary Outcome: Belief of Acupuncture
Description: Patients will be asked "On a scale of 0-10, how much do you believe acupuncture to be a valid treatment for anxiety?" (0=do not believe at all; 10=fully believe)
Time Frame: Up to 30 min post-acupuncture intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Shen Men Acupuncture | Sham Acupuncture | Simulated Acupuncture
Number analyzed (Participants) | 1 | 2 | 1
units on a scale | 8 (0) | 8 (4) | 7 (0)

3. Secondary Outcome: Anxiety Medication Use
Description: Any use of medication use following the acupuncture intervention and before the epidural injection will be documented.
Time Frame: Up to 30 min post-acupuncture intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Shen Men Acupuncture | Sham Acupuncture | Simulated Acupuncture
Number analyzed (Participants) | 1 | 2 | 1
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the duration of the acupuncture intervention (20 minutes).
Arm/Group | Shen Men Acupuncture | Sham Acupuncture | Simulated Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03480919/Prot_SAP_000.pdf